CLINICAL TRIAL: NCT05550675
Title: Prospective Database of Factors Associated With Faecal vs. Double Incontinence in Patients Referred for High Resolution Anorectal Manometry.
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: ProDIM
Record Dates: First submitted 2022-08-12; First posted 2022-09-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Double Incontinence; Faecal Incontinence; Urinary Incontinence
MeSH Terms: conditions — Encopresis; Urinary Incontinence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Double incontinence
  Interventions: Other: Questionnaires
- faecal incontinence
  Interventions: Other: Questionnaires
- controls
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Disease specific questionnaires

SUMMARY:
This study aims to verify the results from our previous retrospective cohort analysis by establishing a database of well-characterised patients prospectively. The different prevalence of neurological disorders, abdominal, urological and obstetrical surgery, diarrhoea and other potential associated factors as well as the importance of abnormalities identified by 3D high resolution anorectal manometry (HARM) will be compared between subjects with feacal incontinence (FI), double incontinence (DI) and controls. Presence and severity of both FI and urinary incontinence (UI) will be evaluated by disease specific questionnaires. Measuring both disease severity and Quality of Life (QoL) is needed to determine the true impact of incontinence. Finally, the impact on quality of life will be compared between both groups.

DETAILED DESCRIPTION:
Double incontinence (DI) is the concomitant incontinence for urine and stool. A 3 - 5 % prevalence among adults has been reported, while 7 - 18 % of community-dwelling adults suffer from faecal incontinence (FI), irrespective of gender. Risk factors for FI include structural anomalies of the anorectal region, disturbed rectal compliance, disturbed anorectal sensation and presence of diarrhoea. Age, body mass index (BMI), obstetrical history (especially parity), anal penetrative intercourse and chronic illness have also been implicated. In contrast, little is known about the pathophysiology of DI. Factors like older age, multiparity, neurological disease and medical comorbidities have been proposed based on analysis from the Nurse's health study. According to our recent retrospective cohort analysis (accepted for publication Acta Gastro-Enterologica Belgica), diarrhoea, neurological disease and previous urological interventions characterise patients suffering from DI. Males most frequently suffer from an underlying neurologic disorder, while anatomical anomalies and urological surgery was more frequently observed in women. There was a trend toward more frequent diarrhoea in both genders. Anorectal manometry parameters could not differentiate between FI alone or DI. However, this result could have been hampered by the use of conventional manometry in contrast to high-resolution 3D manometry.

This study aims to verify the results from our previous retrospective cohort analysis by establishing a database of well-characterised patients prospectively. The different prevalence of neurological disorders, abdominal, urological and obstetrical surgery, diarrhoea and other potential associated factors as well as the importance of abnormalities identified by 3D high resolution anorectal manometry (HARM) will be compared between subjects with FI, DI and controls. Presence and severity of both FI and UI will be evaluated by disease specific questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Self-reported faecal incontinence.

Exclusion Criteria:

* Impossibility to perform the anorectal manometry because of pain, stenosis or organic disease;
* Active (peri)rectal inflammation, including abscess;
* Pregnancy;
* Inability to cooperate during the anorectal manometry
* Impossibility to perform HARM due to pain, stenosis or organic disease;
* Inability to complete the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients referred for HARM for FI are eligible to enroll in the database.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
compose a database of patients suffering from faecal or double incontinence | during inclusion visit
  a database will be created

SECONDARY OUTCOMES:
Confirm the role of diarrhea as a major determinant of double incontinence vs faecal incontinence | during inclusion visit
  this outcome will be assessed using jorge and wexner score
Confirm the role of diarrhea as a major determinant of double incontinence vs faecal incontinence | during inclusion visit
  this outcome will be assessed using vaizey score
Confirm the role of diarrhea as a major determinant of double incontinence vs faecal incontinence | during inclusion visit
  this outcome will be assessed using International consultation on incontinence questionnaire
Confirm the role of diarrhea as a major determinant of double incontinence vs faecal incontinence | during inclusion visit
  this outcome will be assessed using clinical frailty score
Confirm the role of diarrhea as a major determinant of double incontinence vs faecal incontinence | during inclusion visit
  this outcome will be assessed using bristol stool scale
Identify other factors associated with DI vs. FI , | during inclusion visit
  this outcome will be assessed using bristol stool scale
Identify other factors associated with DI vs. FI , | during inclusion visit
  this outcome will be assessed using clinical frailty score
Identify other factors associated with DI vs. FI , | during inclusion visit
  this outcome will be assessed using jorge and wexner score
Identify other factors associated with DI vs. FI , | during inclusion visit
  this outcome will be assessed using vaizey score
Identify other factors associated with DI vs. FI , | during inclusion visit
  this outcome will be assessed using International consultation on incontinence questionnaire
Compare manometric data from HARM in DI vs. FI alone; | during inclusion visit
  this outcome will be assessed using HARM
Assess the prevalence of DI in women and men with FI presenting for HARM; | during inclusion visit
  this outcome will be assessed using HARM
Investigate the impact of UI on the quality of life in DI vs. FI alone. | during inclusion visit
  this outcome will be assessed using the Quality of Life questionnaire (faecal incontinence Quality of Life scale)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No